CLINICAL TRIAL: NCT00901784
Title: Comparative, Randomized, Single Dose, 2-Way Crossover Relative Bioavailability Study of Ranbaxy and Ortho-McNeil Pharmaceutical (Topamax®) 25 mg Topiramate Tablets Following a 50 mg Dose in Healthy Adult Males Under Fasting Conditions
Brief Title: Bioequivalence Study of Topiramate Tablets 25mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 011972
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: Topiramate fasting study
MeSH Terms: interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 25 mg Topiramate tablets of Ranbaxy Laboratories, Ltd
  Interventions: Drug: Topiramate
- 2 (Active Comparator): (Topamax®) 25 mg Topiramate tablets of Ortho-McNeil Pharmaceutical, Inc. New jersey 08869
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — 25mg Tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and Ortho-McNeil Pharmaceutical (Topamax®) 25 mg topiramate tablets following a 50 mg dose under fasting conditions.

DETAILED DESCRIPTION:
This was an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 24 healthy adult male volunteers and 4 alternates. All 28 subjects completed the clinical phase of the study. In each period, subjects were housed from the evening before dosing until after the 24-hour blood draw. Subjects were to return for the 48-, 72-, 96- and 120-hour blood draws. Both periods were separated by a washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. This study involved healthy adult male volunteers, 18-45 years of age, weighing at least 52 kg, who are within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983).
2. Only medically healthy subjects with clinically normal laboratory profiles were enrolled in the study.

Exclusion Criteria:

1. History or presence of significant:

   • cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

   In addition, history or presence of:
   * Hypersensitivity or idiosyncratic reaction to topiramate
   * Nephrolithiasis or gout
   * Alcoholism or drug abuse within the past year
2. Subjects who had been on an abnormal diet (for whatever reason) during the 28 days preceding the study.
3. Subjects who had any drugs or other substances known to be strong inhibitors of CYP (cytochrome P450) enzymes within 10 days of study start.
4. Subjects who had used any drugs or other substances known to be strong inducers of CYP (cytochrome P450) enzymes within 28 days of study start.
5. Subjects who, through completion of the study, would have donated in excess of:

   * 500 mL of blood in 14 days, or
   * 500-750 mL of blood in 14 days (unless approved by the Principal Investigator),
   * 1000 mL of blood in 90 days,
   * 1250 mL of blood in 120 days,
   * 1500 mL of blood in 180 days,
   * 2000 mL of blood in 270 days,
   * 2500 mL of blood in 1 year,
6. Subjects who had participated in another clinical trial within 28 days of study start.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2001-09; Primary Completion 2001-09 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Topiramate 25mg tablets

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharina Services (Clinical Research Center), Saint Laurent, Québec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://www.fda.gov/Safety/Recalls/default.htm
- See also: Related Info — http://www.fda.gov/Safety/MedWatch/default.htm